CLINICAL TRIAL: NCT07392632
Title: MindfulCityU: Implementation and Evaluation of a Mindfulness Mobile Application for Promoting University Students' Mental Health
Brief Title: MindfulCityU-- A Mindfulness Mobile Application for Promoting University Students' Mental Health
Acronym: MindfulCityU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-STA-00001949
Record Dates: First submitted 2026-01-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Depressive Symptoms
Keywords: Digital Mental Health Intervention; Mobile phone application-based; Mindfulness-based Intervention; Depression; Mindfulness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The MindfulCityU provides 8 online modules on mindfulness for participants to access and learn at home through their smartphones and/or computer.
  Participants of waitlist control group participants receive no active intervention at the initial stage and receive the same MindfulCityU at a later stage.
Who Masked: Investigator
Masking Description: A researcher, who is blinded to the randomized allocation of participants and does not involve in the intervention delivery, will do the data collection at before and after the intervention and 2-month follow up. Actually, participants will complete online standardized assessment tools on their intervention outcomes before and after the intervention and 2-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The MindfulCityU provides 8 online modules on mindfulness for participants to access and learn at home through their smartphones and/or computer.
  Interventions: Behavioral: MindfulCityU
- Waitlist Control (Other): The waitlist-controlled group receive standard services from the schools, universities or youth service units.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: MindfulCityU — The MindfulCityU provides 8 online modules on mindfulness for participants to access and learn at home through their smartphones and/or computer. Each participant is expected to complete 8 modules of mindfulness within four weeks, with two sessions released each week to maintain engagement while allowing adequate time for skill development. Beyond the structured curriculum, the application provides daily practice options that accommodate varying time constraints and preferences. These include guided meditations ranging from 5-20 minutes in length, mindful breathing exercises that can be practiced between classes, body awareness practices suitable for dormitory settings, and informal mindfulness reminders integrated throughout the day.
  Arms: Intervention group
Other: Waitlist control — The non-active waitlist-controlled group participants receive standard services from the schools, universities or youth service units. Full access to the digital MBI application is provided following the 4-week waiting period
  Arms: Waitlist Control

SUMMARY:
The research aims to investigate the effectiveness a mobile phone application-based (app-based) mindfulness interventions for university students with mild depressive symptoms.

This study adopts a multicentre randomized control trial two arms research design. A randomised controlled trial will compare a newly designed mobile phone application-based (app-based) mindfulness interventions, named MindfulCityU, with a waitlist control group to determine whether the MindfulCityU produces better intervention outcomes on promoting mental health for university students, including depressive symptoms, mindfulness, and wellbeing. The MindfulCityU provides 8 online modules on mindfulness for participants to access and learn at home through their smartphones and/or computer. Participants of waitlist control group participants receive no active intervention at the initial stage and receive the same MindfulCityU at a later stage.

Participants will complete online standardized assessment tools on their intervention outcomes before and after the intervention and 2-months follow-up. The ethical considerations of this study were reviewed and approved by the Human and Artefacts Ethics Sub-Committee of the City University of Hong Kong in 2025.

DETAILED DESCRIPTION:
University students worldwide face an unprecedented mental health crisis that has intensified significantly in recent years. Meta-analytic evidence demonstrates pooled prevalence rates of 33.6% for depression and 39% for anxiety among this population globally.

In Hong Kong, the mental health crisis among university students is particularly pronounced. Specifically, a longitudinal research conducted between 2016 and 2021 revealed a significant escalation in psychological distress. The study found that 68.5% of students reported diverse depressive symptoms, with 49.4% considered at risk for mental health problems. By 2021, these numbers had escalated dramatically, with depressive symptoms affecting up to 80% of students and at risk cases reaching 60%.

Digital Mindfulness-based Interventions Systematic reviews and meta-analyses provide substantial evidence supporting mindfulness-based interventions (MBIs) for university students. Additionally, mobile phone application-based (app-based) or digital mindfulness interventions have demonstrated particularly promising outcomes among university student populations. It offers several distinct advantages that make them particularly suitable for university populations, including 24/7 accessibility that accommodates irregular student schedules, anonymity that reduces stigma-related barriers to help-seeking, cost-effectiveness that addresses financial constraints common among students, scalability that can reach large numbers of students simultaneously, and personalization capabilities that can adapt to individual needs and preferences.

However, there is a lack of university-specific adaptations in current digital mindfulness interventions. Most existing applications are designed for general adult populations rather than addressing the unique stressors and developmental challenges facing university students, such as academic pressure, social adjustment difficulties, identity development concerns, and career uncertainty.

Research Objective This study aims to addresses these identified gaps by developing and evaluating a culturally adapted, university-specific digital mindfulness intervention, named MindfulCityU. Additionally, this study will examine the mechanisms underlying therapeutic change.

Research Methods This research study adopts mixed methods research design, involving both quantitative and qualitative study. By adopting a randomized controlled trial, the quantitative study aims to investigate the effectiveness of the MindfulCityU on improving mental health for university students. The qualitative study aims to examine the benefits, advantages and limitations of the MindfulCityU from the users' perspective.

Quantitative Research Method

Research Questions and Hypotheses Primary Research Questions RQ1: Does the MindfulCityU intervention improve mental health outcomes (depression, anxiety, stress, well-being) among Hong Kong university students compared to waitlist controls? RQ2: Does app engagement moderate intervention effectiveness, with higher engagement levels predicting greater therapeutic improvements? Secondary Research Questions RQ3: Does baseline mental health symptom severity moderate intervention effectiveness? RQ4: How do participants experience integrating digital mindfulness practices into their daily university routines?

Primary Hypotheses H1 (Primary Effectiveness): Participants receiving the MindfulCityU intervention will demonstrate significantly greater improvements in DASS-Y scores (depression, anxiety, stress) and WHO-5 well-being scores compared to waitlist controls.

H2 (Engagement Moderation): App engagement levels will moderate intervention effectiveness, with higher engagement predicting larger therapeutic gains.

H3 (Baseline Moderation): Baseline symptom severity will moderate intervention effectiveness, with participants having moderate symptoms showing greater improvements than those with mild symptoms.

H4 (Secondary Outcomes): The intervention will produce significant improvements in mindfulness skills (FFMQ-SF), loneliness (UCL-8), and sleep quality (SCI) compared to controls.

Study Design This investigation employs a two-arm randomized controlled trial design to evaluate the efficacy of the MindfulCityU intervention while maintaining scientific rigor and minimizing potential confounding factors. The study design incorporates a 4-week intervention period followed by a 2-month follow-up assessment, allowing for evaluation of both immediate therapeutic effects and sustained benefits over time.

The MindfulCityU application adapted from Professor Daniel Young's established mindfulness curriculum into an interactive digital format specifically adapted for university students and Hong Kong's cultural context. Prior to the main trial implementation, a brief pilot testing phase involving approximately 15 students will be conducted to ensure optimal technical functionality, user experience, and cultural appropriateness.

Power Analysis and Sample Size Justification The sample size calculation is based on previous meta-analytic findings indicating moderate effect sizes for digital mindfulness interventions in university populations. With α = 0.05, power = 0.80, and accounting for an anticipated 20% attrition rate typical in digital intervention studies, the required sample size is 120 participants (60 per group).

Participants and Recruitment The study will recruit 120 CityU students through open promotion and recruitment. Participants will be equal assigned to intervention (n=60) and control (n=60) conditions.

Inclusion criteria (i) current CityU undergraduate or postgraduate students; (2) aged 18-30 years; (3) possess smartphone ownership and reliable internet access necessary for intervention engagement; (4) having mild to moderate depressive symptoms as assessed by the DASS-Y Depression subscale, and a DASS-Y Depression subscale score between 10-23 mild to moderate depressive symptoms; (5) able to listen and read simplified Chinese, Cantonese or English, reflecting Hong Kong's trilingual context.

(6) provide informed consent.

Exclusion criteria:

1. a DASS-Y Depression subscale score above 23 on the DASS-Y Depression subscale, indicating severe symptoms;
2. reporting active suicidal ideation or self-harm behaviors
3. current engagement in psychotherapy or recent medication changes within the previous four weeks;
4. planning to leave the university during the study period.

In particular, participants reporting suicidal ideation, self-harm behaviors or severe depressive symptoms will be immediately referred to crisis intervention services.

Randomization and Blinding Procedures Participants will be randomly allocated to intervention or control conditions using computer-generated randomization sequences with concealed allocation to prevent selection bias. Block randomization will be employed to ensure balanced group sizes throughout the recruitment period. While participants cannot be blinded to their intervention assignment due to the nature of the intervention, outcome assessors will remain blinded to group allocation during data collection and analysis phases to minimize assessment bias.

Intervention Description The MindfulCityU application represents a comprehensive digital mindfulness intervention specifically designed for university students in Hong Kong's cultural context.

The core curriculum consists of eight structured sessions delivered over four weeks, with two sessions released each week to maintain engagement while allowing adequate time for skill development. The first week introduces fundamental mindfulness concepts and practices through Session 1, which covers Introduction to Mindfulness and the Three-Minute Breathing Space technique, and Session 2, which focuses on Body Scan practices and developing physical awareness. These foundational sessions establish basic mindfulness skills and familiarity with core practices.

The second week builds upon foundational skills through Session 3, which introduces Mindful Movement and Stretching practices that integrate physical activity with mindfulness awareness, and Session 4, which teaches the Breathing Space for Difficult Emotions technique, providing practical tools for managing emotional distress. These sessions help participants apply mindfulness skills to common university stressors.

The third week addresses cognitive aspects of mindfulness through Session 5, which focuses on Working with Difficult Thoughts and Feelings, and Session 6, which teaches the concept that Thoughts Are Not Facts through cognitive defusion techniques. These sessions help participants develop a different relationship with negative thinking patterns common among university students.

The fourth week integrates advanced practices through Session 7, which covers Acceptance and Self-Compassion principles particularly relevant for perfectionistic university students, and Session 8, which introduces Loving-Kindness practices and strategies for Maintaining Practice beyond the intervention period.

Beyond the structured curriculum, the application provides daily practice options that include guided meditations ranging from 5-20 minutes in length, mindful breathing exercises that can be practiced between classes, body awareness practices suitable for dormitory settings, and informal mindfulness reminders integrated throughout the day.

Additional features enhance user engagement and safety through progress tracking and streak counters that provide motivational feedback, mood check-ins that enable pattern recognition over time, crisis resources and professional referral pathways for students experiencing severe distress, and integration with CityU counseling services to facilitate seamless transitions to professional care when needed.

Control Condition Waitlist control participants receive access to standard university counselling services and general mental health information emails. Full access to the MindfulCityU application is provided following the 4-week waiting period.

Outcome Assessment Tools.

The primary intervention outcome is improvement in mental health, including depression, anxiety and stress, assessed with the 21-item DASS.

The secondary intervention outcome is improvement in mindfulness, psychological well-being and stress reduction, which are assessed by:

The 20-item Chinese Five Facets Mindfulness Questionnaire Short Form The 8-item UCLA Loneliness Scale (ULS-8) The 8-item Sleep Condition Indicator (SCI) The 5-item Chinese WHO 5-item Well-Being Index (WHO-5)

Data Analysis. An analysis will be performed in accordance with the intent-to-treat principle using multiple imputation method analysis for any missing data. Between group intervention effects will be investigated by using repeated measures of linear mixed model for repeated measures. In the linear mixed model, time, group, and time × group interactions were entered as fixed effects, with a random intercept for the subject. Effect sizes (Hedges' g) are calculated, with values of 0.2, 0.5, and 0.8 considered as small, medium, and large respectively. The predictive values of individual adherence of digital iMBI are analyzed using multiple linear regression analysis, with improved outcome assessment scores as dependent variables.

Qualitative Research Method

Objective. This qualitative study aims to explore the benefits, advantages and limitations of the MindfulCityU from the users' perspective.

Research Design. The qualitative study uses an interpretative interview method with purposive sampling. Semi-structured interviews with 15-20 participants in the current sample will provide rich qualitative data to complement quantitative findings and enhance understanding of intervention effects from participants' perspectives. Each interview will last for 0.5-1 hour. Interview topics will explore intervention experience, perceived benefits and limitations, barriers to engagement, suggested improvements, and integration of mindfulness practices into daily university life. Interviews will be conducted by trained research assistants using standardized interview guides while allowing flexibility to explore emerging themes.

Data collection. Each in-depth interview will be facilitated by a research staff with an interview protocol developed for this study. Participants will be asked questions such as the following: How relevant were the language, examples, and content of today's module of the mindful app to your daily life? How difficult or easy is it to use this app? How often do you use this app? In real life, under what circumstances do you first apply the method you learn from the app? Is there any particular time using the app when you feel "This app really help me"? Do you have any other feedback regarding content, examples, exercises, or app design? The content of the semi-structured in-depth interviews will be audio-recorded and transcribed into verbatim by the research team.

Reflective thematic analysis will be used to identify, analyse and report themes so that themes can be developed both inductively (i.e. data-driven) and deductively (i.e. theory-driven). The research team will systematically read and re-read the transcripts, following the six stages of analysis, including: (1) becoming familiar with the data, (2) generating codes, (3) constructing themes, (4) reviewing potential themes, (5) defining and naming themes, and (6) producing the report. Two research staff compare, review and refine the codes, categories and themes until they reach agreement.

ELIGIBILITY:
Inclusion Criteria:

(i) current undergraduate or postgraduate students; (ii) aged 18-30 years; (iii) possessing smartphone ownership and reliable internet access necessary for intervention engagement; (iv) having a score between 10-23 on the DASS-Y Depression subscale indicating a mild to moderate depressive symptom; and (v) provide informed consent

Exclusion Criteria:

(i) students currently engaged in formal mindfulness training exceeding one session per week will be excluded to prevent confounding effects from concurrent mindfulness practice; (ii) those scoring above 23 on the DASS-Y Depression subscale, indicating severe symptoms, will be excluded and referred to appropriate clinical services to ensure their safety and access to needed care; (iii) students reporting active suicidal ideation or self-harm behaviors will be immediately referred to crisis intervention services and excluded from study participation to prioritize their safety; (iv) current engagement in psychotherapy or recent medication changes within the previous four weeks; (v) students planning to leave the university during the study period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Chinese Depression Anxiety Stress Scale Youth Version (DASS-Y) | This scale will be used at baseline, the 5th week, and the 13rd week.
  The primary intervention outcome is improvement in mental health, including depression, anxiety and stress, assessed with the 21-item DASS-Y which has been demonstrated good validity and reliability (α = 0.80 for anxiety subscale, 0.83 for depression subscale, 0.82 for stress subscale, and 0.92 for whole scale; Cao et al., 2023). Each item (e.g. I felt down-hearted and blue) is scored from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The scores are summed over the items with higher scores indicating a higher severity of symptoms

SECONDARY OUTCOMES:
Chinese Five Facets Mindfulness Questionnaire Short Form (FFMQ) | This scale will be used at baseline, the 5th week, and the 13rd week.
  The Chinese Five Facets Mindfulness Questionnaire Short Form (FFMQ; Fong et al., 2021), which is a 20-item scale with good validity and internal consistency (Cronbach's α range from 0.77 to 0.85), was used to assess participants' level of mindfulness. Each item (e.g., "I pay attention to sensations, such as the wind in my hair or sun on my face") is rated on a 5-point Likert scale (1 = Never or very rarely true; 5 = Very often or always true). A higher score indicates a higher level of mindfulness
UCLA Loneliness Scale (ULS-8) | The scale will be used at baseline, the 5th week, and the 13rd week.
  The UCLA Loneliness Scale (ULS-8), which is an 8-item scale with good validity and internal consistency (Cronbach's α = 0.80), is used to assess perceived loneliness (Xu et al., 2018). Each item (e.g., feel that a lack of companionship) is rated on a 4-point Likert-type scale ranging from 0 to 4. A higher score indicates a higher level of perceived loneliness
Sleep Condition Indicator (SCI) | The scale will be used at baseline, the 5th week, and the 13rd week.
  The Sleep Condition Indicator (SCI), which is an 8-item scale with good validity and internal consistency (Cronbach's α = 0.82), is used to assess perceived loneliness (Meng et al., 2022). Each item (e.g., how would you rate your sleep quality?) is rated on a 5-point Likert-type scale ranging from 1 (never) to 4 (always). A higher score indicates a better sleep quality over the last month (Meng et al., 2022).
Chinese WHO 5-item Well-Being Index (WHO-5) | The scale will be used at baseline, the 5th week, and the 13rd week.
  The Chinese WHO 5-item Well-Being Index (WHO-5) is a 5-item scale for assessing subjective well-being with satisfactory validity and internal consistency (Cronbach's α = 0.85; Fung et al., 2022). Each item (e.g., I have felt calm and relaxed) is rated on a 6-point Likert-type scale ranging from 0 (at no time) to 5 (all of the time). A higher score indicates a better well-being

CONTACTS AND LOCATIONS:
Locations (1):
- City University of Hong Kong, Kowloon Tong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oei TP, Sawang S, Goh YW, Mukhtar F. Using the Depression Anxiety Stress Scale 21 (DASS-21) across cultures. Int J Psychol. 2013;48(6):1018-29. doi: 10.1080/00207594.2012.755535. Epub 2013 Feb 21. PMID 23425257
- [Background] Xu S, Qiu D, Hahne J, Zhao M, Hu M. Psychometric properties of the short-form UCLA Loneliness Scale (ULS-8) among Chinese adolescents. Medicine (Baltimore). 2018 Sep;97(38):e12373. doi: 10.1097/MD.0000000000012373. PMID 30235699
- [Background] Philippe TJ, Sikder N, Jackson A, Koblanski ME, Liow E, Pilarinos A, Vasarhelyi K. Digital Health Interventions for Delivery of Mental Health Care: Systematic and Comprehensive Meta-Review. JMIR Ment Health. 2022 May 12;9(5):e35159. doi: 10.2196/35159. PMID 35551058
- [Background] Pan, Y., Li, F., Liang, H., Shen, X., Bing, Z., Cheng, L., & Dong, Y. (2024). Effectiveness of Mindfulness-Based Stress Reduction on Mental Health and Psychological Quality of Life among University Students: A GRADE-Assessed Systematic Review. Evidence-Based Complementary and Alternative Medicine : eCAM, 2024, 8872685. https://doi.org/10.1155/2024/8872685
- [Background] Linardon J, Torous J, Firth J, Cuijpers P, Messer M, Fuller-Tyszkiewicz M. Current evidence on the efficacy of mental health smartphone apps for symptoms of depression and anxiety. A meta-analysis of 176 randomized controlled trials. World Psychiatry. 2024 Feb;23(1):139-149. doi: 10.1002/wps.21183. PMID 38214614
- [Background] Li, W., Zhao, Z., Chen, D., Peng, Y., & Lu, Z. (2022). Prevalence and associated factors of depression and anxiety symptoms among college students: A systematic review and meta-analysis. Journal of Child Psychology and Psychiatry, and Allied Disciplines, 63(11), 1222-1230. https://doi.org/10.1111/jcpp.13606
- [Background] Fung, S., Kong, C. Y. W., Liu, Y., Huang, Q., Xiong, Z., Jiang, Z., Zhu, F., Chen, Z., Sun, K., Zhao, H., & Yu, P. (2022). Validity and Psychometric Evaluation of the Chinese Version of the 5-Item WHO Well-Being Index. Frontiers in Public Health, 10. https://doi.org/10.3389/fpubh.2022.872436
- [Background] Fong TCT, Wan AHY, Wong VPY, Ho RTH. Psychometric properties of the Chinese version of Five Facet Mindfulness Questionnaire-short form in cancer patients: a Bayesian structural equation modeling approach. Health Qual Life Outcomes. 2021 Feb 10;19(1):51. doi: 10.1186/s12955-021-01692-1. PMID 33568146
- [Background] Cao, C., Liao, X., Gamble, J. H., Li, L., Jiang, X.-Y., Li, X.-D., Griffiths, M. D., Chen, I.-H., & Lin, C.-Y. (2023). Evaluating the psychometric properties of the Chinese Depression Anxiety Stress Scale for Youth (DASS-Y) and DASS-21. Child and Adolescent Psychiatry and Mental Health, 17(1), 106. https://doi.org/10.1186/s13034-023-00655-2